CLINICAL TRIAL: NCT00670904
Title: Randomized Trial Assessing the Effectiveness of a Pharmacist-Delivered Program for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Collaborators: Prevent Cancer Foundation (Other)
Responsible Party: Larry A. Dent, The University of Montana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M29670
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2008-04

CONDITIONS: Tobacco Use Disorder; Smoking
Keywords: Smoking cessation; Pharmacist-delivered
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Pharmacist-delivered group program for smoking cession.
  Interventions: Other: Pharmacist-delivered group program for smoking cessation
- 2 (Placebo Comparator): Brief standard care session for tobacco smoking cessation delivered over the telephone.
  Interventions: Other: Brief standard care session for smoking cessation delivered over the telephone

INTERVENTIONS:
Other: Pharmacist-delivered group program for smoking cessation — Participants assigned to the treatment group participated in a pharmacist-delivered program at the clinic. The six-hour program consisted of three in-person sessions delivered at 2-week intervals over 5 weeks to a small group of smokers. Participants were offered their choice of one medication either bupropion IR or nicotine patch using doses and durations based on current medical practices. Participants receiving bupropion received a quantity sufficient to complete 12 weeks of therapy. Participants receiving nicotine patches received a quantity sufficient to complete 8 weeks of step-down therapy.
  Arms: 1
Other: Brief standard care session for smoking cessation delivered over the telephone — Those assigned to the control group received one 5 to 10 minute session delivered by the clinical pharmacist over the telephone that included all the components of standard care recommended by the Clinical Practice Guidelines for brief interventions delivered by health care providers. Participants were offered their choice of one medication either bupropion IR or nicotine patch using doses and durations based on current medical practices. Participants receiving bupropion received a quantity sufficient to complete 12 weeks of therapy. Participants receiving nicotine patches received a quantity sufficient to complete 8 weeks of step-down therapy.
  Arms: 2

SUMMARY:
This randomized trial compared the effectiveness of a three session pharmacist-delivered group program for smoking versus one 5 to 10 minute standard care session delivered over the telephone on 7-day point prevalence quit rates. Participants in both groups were offered their choice of bupropion IR or nicotine patch at no cost. At 6 months after the established quit date, self-reported cessation was biochemically verified using tests for urinary cotinine.

ELIGIBILITY:
Inclusion Criteria:

* Smoked one or more cigarettes daily for 7 days
* Somewhat ready to quit in the next 2 weeks (4 or more on a 10- point scale)
* Willing and capable of attending three scheduled sessions at the clinic
* Interested in participating in the study

Exclusion Criteria:

* Planned to leave the area in the next 6 months
* Used pharmacotherapy for smoking cessation in the last 30 days
* Used other forms of tobacco in the last 30 days
* Schizophrenia
* Prior participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2005-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable for the study was biochemically verified 7-day point prevalence smoking cessation at 6 months, defined as having smoked no cigarettes - not even a puff - for the previous 7 days. | 6 months

SECONDARY OUTCOMES:
Secondary outcomes included 30-day point prevalence abstinence and prolonged abstinence (>6 months). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Larry A. Dent, Pharm.D., Principal Investigator — The University of Montana
Locations (1):
- Missoula VA Clinic, Missoula, Montana, United States